CLINICAL TRIAL: NCT02203006
Title: Constitution of an Open Monocentric Cohort of HIV Infected Patients
Brief Title: HIV Patients Cohort
Acronym: OVIHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IDRCB : 2010-A00417-32
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Patients Affected by the HIV
Keywords: HIV,; infection,; cohort
MeSH Terms: conditions — Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OVIHD (Other): Cohort and a blood sample collection will be done with data and blood of HIV infected patients
  Interventions: Biological: OVIHD

INTERVENTIONS:
Biological: OVIHD — 7 ml of blood will be taken during a follow-up consultation and kept in a biological collection. Clinical data will be collected in a database.
  Other Names: Blood sample

SUMMARY:
The purpose of this study is to improve our knowledge concerning HIV infection, treated or not, in the current conditions of care to optimize it.

DETAILED DESCRIPTION:
Since the arrival of highly active tritherapies, HIV infection became mainly an ambulatory chronic pathology centred on a long term care taking into account the complication of long-term treatment as well as the arisen of new problem bound to a prolonged survival and ageing. So the care is more and more in a prevention and screening approach with in particular the care of metabolic and cardiovascular complication due to antiretroviral treatment.

As a reorganization of the coverage of the HIV infected people take place on the Hotel Dieu Hospital it thus seems important to double this care optimization with a clinical research side. This will be done in constituting an HIV patient cohort including a blood sample collection to contribute to the vigilance of the complication to due the infection.

Our ultimate objective is to optimize the selection of the treatment. It is important to do it to be able to have, on many years duration, precise clinical information and biological sample allowing to realize later some assay and analyse the influence of some genetic markers.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old,
* Patients with an HIV infection
* patients having given their written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1613 (Actual)
Dates: Start 2011-10-19 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
HIV infection | 10 years
  The HIV cohort will be constituted in collecting cardiovascular, neurological clinical data and medical past history (in case of women patient)

SECONDARY OUTCOMES:
Comorbidity and complication in HIV infected patients | 10 years
  The HIV cohort will be constituted in collecting cardiovascular, neurological clinical data and medical past history (in case of women patient)
efficiency of the current antiretroviral therapeutic diets | 10 years
  The HIV cohort will be constituted in collecting cardiovascular, neurological clinical data and medical past history (in case of women patient)
Blood sample collection | 10 years
  To put in relation the clinical-biological relevant biological or genetic data of the follow-up a blood sample will be constituted. 7 ml will be taken to each patient and kept in a collection

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Tréluyer, MD, PhD, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Hôtel Dieu, Paris, France